CLINICAL TRIAL: NCT06188312
Title: Main Occupational Health Hazards Among Workers Of Superphosphate Fertilizer Factory in Assiut and Evaluation of a Health Education Program On Dangers of Respirable Chemicals.
Brief Title: Occupational Hazards Among Workers of Superphosphate Fertilizer Factory
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Israa salah El-Din Shaker, Assistant Lecturer, Assiut University
Other Study IDs: Israa.S.Shaker
Record Dates: First submitted 2023-12-18; First posted 2024-01-03 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Occupational Exposure; Health Knowledge, Attitudes, Practice
Keywords: superphosphate factory; Health hazards; Health education
MeSH Terms: conditions — Behavior; Health Education

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Health education program — A pretest questionnaire will be filled out, asking the participants about their knowledge, attitudes, and practices toward chemical hazards and the use of personal protective equipment (PPE) then analysis of the obtained pre-test data will be done.
  we will apply a health education program. Development phase: developing the message of the health education program and preparing the materials (slide presentation, brochures, and an educational video).Implementation phase: A group health education session through face-to-face, one hour long, interactive lecture combined with slide presentation will be carried out by the researcher. Evaluation phase: A post-test will be done, after 6 months of the first session, to assess the changes of their knowledge and attitude after the intervention.

SUMMARY:
The study aims:

* To identify the main occupational health hazards to which the superphosphate fertilizer industry workers are exposed.
* To identify the respiratory and auditory health effects of these hazards and associated risk factors among those workers.
* To clarify the knowledge, attitudes, and practices of workers towards the chemical health hazards affecting the respiratory system (dust and hazardous gases).
* To assess the effect of health education program on workers' knowledge, attitudes, and practices towards these hazards and the use of personal protective equipment (PPE).

DETAILED DESCRIPTION:
Fertilizers are compounds that provide nutrients to plants to increase and maintain maximum crop yield. They are classified as organic, inorganic, or chemical fertilizers. Organic fertilizers are by-products of livestock, fish, and food. Chemical fertilizers (CFs) are manufactured using different proportions of major and minor chemical nutrients. Although the use of fertilizers in the agricultural sector is inevitable to meet increasing food demand, the production of fertilizers and by-products poses health and safety challenges. Two basic types of fertilizers are produced by Egyptian companies, which include nitrogenous and phosphate fertilizers (PF). Normal superphosphate (NSP) is manufactured from the reaction between phosphate rocks (PR) and sulfuric acid. There are some side chemical reactions involving fluorine and silica of PR producing H2SiF6 (fluorosilicic acid) and other hydrogen fluorides. PF industry is one of the most environmentally polluting industries in Egypt. Workers in the PF industry are exposed to many chemical and physical hazards. Hazardous gas emissions include gaseous fluorides in the form of hydrofluoric acid (HF) and silicon tetrafluoride (SiF4), and sulfur dioxide (SO2). SO2 is one of the five major air pollutants in the world . It is an irritant gas that causes changes in the mechanical functions of the upper airways of the lung, resulting in bronchitis, and bronchoconstriction. Sulfuric acid mists also irritate the human airways causing pulmonary epithelium damage. Chronic fluoride exposure is characterized by accumulation mainly in hard tissues such as teeth and bones in the form of bone deformities (skeletal fluorosis) and dental mottling (dental fluorosis), and non-skeletal fluorosis (other system manifestations such as respiratory manifestations such as asthma. In Egypt, a descriptive study was conducted on 180 exposed workers in a phosphate fertilizer factory at Kafr El-Zayat City, revealed that self-reported respiratory manifestations were found in 74/180 workers (41.11%) and abnormal ventilatory functions were confirmed in (43/180, 23.9%) with a prominence of the obstructive pattern . Noise is one of the most important physical hazards in the fertilizer industry that has become a major problem in all industrial sectors. An unmatched case-control study was carried out among fertilizer factory workers in Malaysia, revealed that cases were at 3.5 times greater risk of being exposed to more than 85 dB compared to the control. There is a lack of published research assessing the occupational health problems among workers in the phosphate fertilizer industry in Upper Egypt and especially in Assiut.

ELIGIBILITY:
Inclusion Criteria:

All workers in the superphosphate fertilizer factory with a duration of work more than one year.

Exclusion Criteria:

* Workers who had history of any chronic respiratory diseases before employment, and those who had history of hearing loss before employment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Phase one(survey): The total number of workers in the factory is 660.They were classified according to the levels of exposure to high exposure (including the production and engineering sectors) and low exposure (including the administrative sector).
  * The high exposure group represented 76 % of workers [58% (380 workers) of the production workers and 18% (120 workers) of the engineering sector].
  * The low exposure group represented 24% (160 workers) of the administrative sector.
Sampling Method: Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
prevalence of respiratory and auditory problems among workers of the superphosphate fertilizer factory. | 1-1-2024 to 1-6-2024
  percentage of workers who had respiratory and auditory affection

SECONDARY OUTCOMES:
Mean score difference of knowledge, attitudes, and practices before and after the health education program among workers of the superphosphate fertilizer factory. | 1-6-2024 to 1-12-2024
  mean difference of knowledge, attitudes, and practicesof the workers before and after application of the health education program

CONTACTS AND LOCATIONS:
Overall Officials: Israa Salah El Din, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chien, S. H., Prochnow, L. I. & Cantarella, H. (2009) Chapter 8 Recent Developments of Fertilizer Production and Use to Improve Nutrient Efficiency and Minimize Environmental Impacts, Advances in AgronomyAcademic Press, 267-322.
- [Background] Zayed HA, Salah N, Hassan NM, Elmagid DA. Assessment of respiratory health and environmental safety measures in phosphate fertilizer industry in the middle region of the Nile Delta, Egypt. Environ Sci Pollut Res Int. 2020 Oct;27(28):35008-35016. doi: 10.1007/s11356-020-09817-7. Epub 2020 Jun 25. PMID 32583121
- [Background] Huda, N. U. & Territory, I. C. (2022) REVIEW ON OCCUPATIONAL HEALTH AND SAFETY ISSUES IN FERTILIZER INDUSTRY.
- [Background] Saffree Jeffree M, Ismail N, Awang Lukman K. Hearing impairment and contributing factors among fertilizer factory workers. J Occup Health. 2016 Sep 30;58(5):434-443. doi: 10.1539/joh.16-0043-OA. Epub 2016 Aug 4. PMID 27488035
- [Background] Komarnisky LA, Christopherson RJ, Basu TK. Sulfur: its clinical and toxicologic aspects. Nutrition. 2003 Jan;19(1):54-61. doi: 10.1016/s0899-9007(02)00833-x. PMID 12507640
- [Background] Leikam, D. F. & Achorn, F. P. (2005) Phosphate fertilizers: production, characteristics, and technologies. Phosphorus: Agriculture and the environment, 46, 23-50.
- [Background] Geravandi, S., Goudarzi, G., Babaei, A. A., Takdastan, A., Mohammadi, M. J., Niri, M. V., Salmanzadeh, S. & Shirbeigi, E. (2015) Health endpoint attributed to sulfur dioxide air pollutants. Jundishapur Journal of Health Sciences, 7(3).
- See also: Elessent Clean Technologies (2023) Sulfuric Acid in the Phosphate Fertilizer Industry, 2023 — https://elessentct.com/industries/phosphate-fertilizer/